CLINICAL TRIAL: NCT04789265
Title: Instrumental Soft Tissue Mobilization in Patients With Chronic Neck Pain: a Randomized Controlled Trial
Brief Title: Instrumental Soft Tissue Mobilization in Patients With Chronic Neck Pain
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Ayşegül BOSTAN (Other)
Responsible Party: Sponsor-Investigator, Ayşegül BOSTAN, physiotherapist, research assistant, Medipol University
Organization: Medipol University (Other)
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 10376522
Record Dates: First submitted 2021-03-02; First posted 2021-03-09 (Actual); Last update posted 2021-05-26 (Actual); Status verified 2021-05

CONDITIONS: Neck Pain
MeSH Terms: conditions — Neck Pain

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Combined Therapy (Instrumented Soft Tissue Mobilization) (Experimental)
  Interventions: Other: instrumented- assisted soft tissue mobilization (IASTM)
- Control Group (Exercise Therapy) (No Intervention)

INTERVENTIONS:
Other: instrumented- assisted soft tissue mobilization (IASTM) — IASTM is a new, non-invasive, conservative therapeutic approach. Instead of the therapist's hands and fingers in treatment, these devices are used to provide contact mobilization power. AYDM intervention, such as friction, rubbing massage treatments, requires the therapist to apply a significant amount of pressure. The main purpose of IASTM is to eliminate scar tissue and to restore the normal function of the tissue following soft tissue regeneration.
  Arms: Combined Therapy (Instrumented Soft Tissue Mobilization)

SUMMARY:
In this study, it was planned to investigate the effectiveness of instrument-assisted soft tissue mobilisation (IASTM) in patients with chronic neck pain. Forty eight individuals with chronic neck pain between the ages of 18-70 were included in the study. Individuals were randomly divided into two groups as Combined Therapy (CT) (n = 24) and Exercise Therapy (ET) (n = 24) groups. All exercises were applied to the participants for 4 weeks, 3 times a week, by an experienced physiotherapist for 5 years under supervision. ET which included stretching and strengthening exercises involving the neck, shoulder and around the scapula muscles applied according to the tolerance of the individuals and targeted to be most beneficial in daily life activities.

CT in addition to the ET applied 3 times a week for 4 weeks, the participants received a total of 8 sessions of IASTM on the days they came to the treatment twice a week, before the ET. As soon as the participants came to the session, IASTM was applied first. Following the IASTM application, ET was applied in the same protocol and under the same therapist supervise with the ET group.

Before and after treatment, deep neck flexor muscle endurance (DNFME), pain severity with Visual Analogue Scale (VAS) and Brief Pain Inventory (BPI), functional status with Neck Disability Index (NDI), quality of life with Nottingham Health Profile (NHP) treatment and treatment satisfaction was evaluated.

ELIGIBILITY:
Inclusion Criteria, Exclusion Criteria:

Individuals aged 18-70 years with neck pain due to a nonspecific disorder for at least 3 months were included.

Individuals with history of cancer (within the last five years), pregnancy, serious skin disorders, previous neck surgery, disc prolapse, spondylolisthesis, vertebral fractures, spinal stenosis, arthritis, osteoporosis, recent neck trauma (within the last 48 hours), severe night pain, symptoms of infection, psychological disorder, and those who received therapy for neck pain in the last 6 months were not included.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 48 (Actual)
Dates: Start 2020-06-26 (Actual); Primary Completion 2020-10-05 (Actual); Study Completion 2020-12-11 (Actual)

PRIMARY OUTCOMES:
Neck Flexor Muscle Endurance | baseline to 4 weeks after
  Neck flexor endurance of the participants were evaluated with a stopwatch for holding their neck in lying position.

SECONDARY OUTCOMES:
Nottingham Health Profile | baseline to 4 weeks after
  NSP is a general health status questionnaire that measures the physical, emotional and social conditions of individuals. The questionnaire consists of 38 items and 6 sub-sections: physical mobility (8 items), pain (8 items), sleep (5 items), emotional reactions (9 items), social isolation (5 items) and energy level (3 items). consists of. Each item is answered as "yes" or "no". The score that can be obtained from each section varies between 0 and 100.
Neck Disability İndex | baseline to 4 weeks after
  The index, which evaluates subjective symptoms and activities of daily living, consists of 10 parts (pain intensity, personal care, lifting, reading, headache, concentration, work life, driving, sleep and leisure activities). There are 6 options ranging from 0 to 5 points for each section. The total score ranges from 0 to 50 (0: no apology; 50: maximum disability), with a higher total score indicating an increased disability.
Visual Analog Scale | baseline to 4 weeks after
  This scale consists of a 10 cm linear line. The starting point of the line is 0, no pain; the last point, 10, the most severe pain encountered in life; 5 means a moderate pain. The subjects were asked to rate the severity of their pain numerically on the scale.

CONTACTS AND LOCATIONS:
Locations (1):
- Aysegul Bostan, Istanbul, Beykoz, Turkey (Türkiye)